CLINICAL TRIAL: NCT05982132
Title: Weight Changes Among Martinican Prisoners
Acronym: NUTRI-LAJÔL
Status: Recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 19_RIPH3_13
Record Dates: First submitted 2022-11-14; First posted 2023-08-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Weight Gain; Weight Loss
Keywords: Prisoners; Body weight; Male; French West Indies; Epidemiology
MeSH Terms: conditions — Weight Gain; Weight Loss; Body Weight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: anthropometric measurement — Measurement of weight and other anthropometrics data

SUMMARY:
Assessment of body weight change among prisoners in Martinique between admission in jail and 3 months later expressed as a percentage of admission weight. Intensity of physical activities, nutrition intakes and psychological state are also studied to describe associated factors to body weight change.

DETAILED DESCRIPTION:
Several studies described how weight of prisoners may vary during incarceration. Taking or losing weight both have health consequences but are also a warning signal for several pathologies. Female prisoners are more likely getting fat, data are rare and contradictory about male prisoners. A single study was conducted in mainland France and including few men. Furthermore, Martinique is a department where the prevalence of overweight and diabetes in the general population are higher than the national average. Prisoners most often have socio-demographic featuring and morbidity different from the general population (more men, some over-represented age groups, addictive behaviors and more frequent mental health problems ...). Aspects nutritional information is less often documented. What about the weight variation of people held in Martinique? Is incarceration always accompanied by weight gain? What are factors associated with weight variation? This study aims to answer to those questions by including all men newly admit in the only martinican jail aged from 18 to 44 years and consenting. During admission medical consultation, prisoners will fill guided by the investigator doctor of self-questionnaires of the evaluation of the level of physical activity, assessment of nutritional intakes and psychological state before incarceration. Measurement of weight and other anthropometrics data will be done, investigator doctor will collect data about socio-economic featuring, medical history and treatment. Three months later, a research technician will interview included prisoners in their life place and guide them to fill new self-questionnaires of the evaluation of the level of physical activity, assessment of nutritional intakes and psychological state during incarceration. Measure weight and other anthropometrics data and collecting data about new treatment, stopping tobacco will be done during this interview.

ELIGIBILITY:
Inclusion Criteria:

* all men newly incarcerated in martinican jail during inclusion period
* age between 18 and 44 years old
* having given his consent

Exclusion Criteria:

* female
* 44 years old and up
* not understanding or speaking French or English

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is based on gender : only men
Study Population: all men aged from 18 to 44 incarcerated in martinican jail during inclusion period and consenting
Sampling Method: Probability Sample
Enrollment: 227 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Weight change between baseline and Month 3 visit among men aged 18 to 44, newly incarcerated in martinican jail | The primary outcome will be collected at baseline (entrance medical examination) and Month 3 visit
  Weight change between baseline and Month 3 visit expressed as a percentage

SECONDARY OUTCOMES:
Body mass index measurement change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and Month 3 visit
  BMI in kg/m^2
Waist size measurement change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and visit at 3 months
  Waist size in centimeters
Lean mass measurement change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and visit at 3 months
  Lean body mass is measured with a body composition scale in kg
Body fat measurement change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and visit at 3 months
  Body fat is measured with a body composition scale in percentage
Percentage body water measurement change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and visit at 3 months
  Percentage body water is measured with a body composition scale
Visceral fat measurement change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and visit at 3 months
  Visceral fat is measured with a body composition scale in level
Basal metabolic rate measurement change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and visit at 3 months
  Basal metabolic rate is measured with a body composition scale in kCal
Sportive activities intensity change can be associated with weight change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and visit at 3 months
  Change in intensity of sports activities measured using a self-questionnaire according to RICCI & GAGNON
The variation of nutrition intakes change can be associated with weight change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and visit at 3 months
  The variation in nutritional intake is assessed by means of a questionnaire
Psychological state change can be associated with weight change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and visit at 3 months
  Change in psychological state will be assessed by the STAY self-questionnaire
New treatment can be associated with weight change between baseline and Month 3 visit | This outcome will be collected at baseline (entrance medical examination) and visit at 3 months
  Introduction or not of new treatment that may have an impact on the weight per data collection. Name of new treatment (in case of) will be notifed in order to search if weigth change is one of his sides effect known.

CONTACTS AND LOCATIONS:
Overall Officials: Anaïs BOURGUIGNON D'HERBIGNY, MD, Principal Investigator — Martinique University Hospital Center
Locations (1):
- CHU Martinique, Ducos, Martinique

IPD SHARING:
Plan to Share IPD: No